CLINICAL TRIAL: NCT06573034
Title: Standing Like a Tree: Effects and Mechanisms of Daoist Zhanzhuang on Human Flourishing
Brief Title: Daoist Zhanzhuang and Human Flourishing
Acronym: Z-Flo
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Charlotte (Other)
Responsible Party: Principal Investigator, Zhuo Job Chen, Associate Professor, University of North Carolina, Charlotte
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB-24-0749; 32539 (Other Grant/Funding Number: Templeton World Charity Foundation)
Record Dates: First submitted 2024-08-23; First posted 2024-08-27 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-08

CONDITIONS: Stress, Physiological; Stress, Psychological; Inflammatory Response; Well-Being, Psychological
Keywords: Human Flourishing; Daoist Zhanzhuang (Chan Chuang); Heart Rate Variability; Immune Function; Mysticism
MeSH Terms: conditions — Stress, Psychological; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: The two arms will include an active control condition (i.e., sham wall squat) and the Daoist Zhanzhuang condition.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be kept unaware of both their assigned condition and the study hypotheses. The research staff responsible for conducting the intervention and assessments will be blinded to the study hypotheses.Different researchers will be assigned to handle the procedures of recruitment, intervention, data collection, and analyses. Outcome assessors and data managers will not participate in participants' screening and allocation, and outcome assessors will maintain blindness to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Daoist Zhanzhuang (Experimental): Individuals in this condition will learn and maintain the Zhanzhuang posture, endorsed by this study's religious practitioner and validated by two independent Daoist experts. The core posture involves: a) Standing with feet shoulder-width apart, knees slightly bent, and toes pointed forward; b) Opening the hips slightly to the side as if holding a ball between the legs; c) Sitting slightly back and tucking in the abdomen and tailbone; d) Keeping the back straight while holding in the chest; e) Raising the arms to a height over the chest but under the shoulders as if embracing a tree trunk; f) Facing palms toward the body with fingers apart as if holding a ball; g) Relaxing the shoulders and lowering the elbows in a stationary stance; h) Pointing the head upward as if balancing an object on top of the head; i) Tucking in the chin; j) Breathing naturally, with a focus on the lower abdominal area.
  Interventions: Behavioral: Daoist Zhanzhuang
- Sham Wall Squat (Active Comparator): Individuals in this condition will be directed to perform a sham wall squat, essentially a prescribed way to stand straight leaning against the wall. Key instructions include: a) Standing tall with the head and back resting against the wall; b) Positioning feet shoulder-width apart and a foot away from the wall; c) Slightly bending and engaging leg muscles; d) Relaxing hands on the side of the body; e) Concentrating on the balance of weight.
  Interventions: Behavioral: Sham Wall Squat

INTERVENTIONS:
Behavioral: Daoist Zhanzhuang — Each session of practice will last 30 minutes, and participants are expected to participate every day for 3 months. During the initial 3 weeks, participants will engage in in-person sessions 3 times a week. On non-session days, they can choose to either attend a Zoom practice session with the coach or submit a recording of their individual practice for fidelity check. In Week 4, participants will attend an in-person session for both practice and assessment. Over the subsequent 8 weeks, participants will either attend in-person or Zoom sessions, with a total of 3 check-in sessions.
  Arms: Daoist Zhanzhuang
Behavioral: Sham Wall Squat — Same as the Zhanzhuang group.
  Arms: Sham Wall Squat

SUMMARY:
This project investigates the impact of Daoist Zhanzhuang (sometimes spelled as Chan Chuang) on human flourishing, and explores the physiological, psychological, and spiritual mechanisms. This study will be a two-arm randomized controlled trial, with mixed-methods and repeated-measures assessment of outcome variables. The two arms will include an active control condition (i.e., sham wall squat) and the Daoist Zhanzhuang condition. Outcome variables will include physiological measures of heart rate variability and inflammatory biomarkers, psychological scales of human flourishing variables, phenomenological interviews of mystical experiences, and daily ecological momentary assessment of human flourishing and mysticism. Randomly assigned into two conditions, 120 participants will complete a three-week intensive practice phase with 9 in-person sessions, followed by a nine-week self-guided practice phase with 4 in-person check-in sessions, and 3 follow-up practice and assessment sessions. Complete assessment (physiological measures, psychological scales, and phenomenological interviews) will be administered at five time points: T1 at about two weeks before the intervention, T2 at the end of the three-week intensive practice, T3 at the end of the 3-month intervention, T4 at the 6-month follow-up, and T5 at the 12-month follow-up. In addition, daily ecological momentary assessment of flourishing variables and practice-induced experiences will be administered daily after the practice for the entire 3-month intervention period.

DETAILED DESCRIPTION:
Zhanzhuang, "standing like a tree," is a standing meditation rooted in Daoism, with its earliest form documented on a Chinese silk manuscript called Daoyintu, dating back two thousand years. By aligning the human body, Zhanzhuang promotes the circulation and accumulation of qi, fostering enhanced energy, health, and healing. In Daoist theology, qi acts as an intermediary connecting physical energy (jing) and the spirit (shen). Zhanzhuang serves as a foundational practice that establishes conditions for the convergence of the physical and non-physical aspects of human being. One of the greatest Daoist spiritual achievements lies not in transcending the body but in the harmonious integration of body and spirit. While many definitions of spirituality emphasize transcendence and non-physicality, the study of Zhanzhuang suggests that immanence and embodiment are equally significant in defining spirituality.

Data from eight clinical trials demonstrate that Zhanzhuang can improve physical endurance, reduce fatigue, enhance body awareness and emotional regulation, and promote better quality of life. However, none of the studies included an active control group, so it is difficult to dissect the effects from merely extra exercise. Overall, existing studies have construed Zhanzhuang (or more generally qigong) as an out-of-the-box alternative behavioral medicine approach, without trying to understand why and how it works. None have examined its spiritual underpinnings. This decontextualized scholarly work can be a disservice to both the Daoist community, where Zhanzhuang practice originates and is taught, and to the public they serve. Zhanzhuang could offer more than being another complementary therapy. Among many benefits, the practice shows that there is a spiritual aspect that resides within one's physical body, and the spirit and the body can join each other to make genuine flourishing possible.

In addition to documenting the effects of Zhanzhuang on human flourishing, the current study will show why and how Zhanzhuang works. Primary hypotheses posit that Zhanzhuang fosters enhanced energy, resilience, and healing. These effects will be evidenced through physiological changes, such as increased parasympathetic activity and improved immune functioning, as well as psychological responses, including elevated vitality, enhanced stress coping abilities, and overall well-being. These effects may be partially attributed to an augmented interoceptive awareness and a deepened psychological insight into previously avoided emotions. Furthermore, the study explores the potential moderation of these effects by acquired mystical experiences, serving as indicators of spiritual progress within the practice of Zhanzhuang. Lastly, the research will delve into the trajectory of change and within-subject causal processes, examining the relationship between mystical experiences and human flourishing over the 3-month practice period through intensive longitudinal measures.

ELIGIBILITY:
Inclusion Criteria:

1. young adults aged between 18 and 25 years old when they enroll;
2. be willing and available (e.g., intend to remain in Charlotte or the surrounding area or willing to travel to UNCC campus for in person visits) to participate to 12 month study;
3. able to stand for 30 minutes;
4. scoring above 18 on the Perceived Stress Scale (moderate stress); and
5. able to read, speak and understand English.

Exclusion Criteria:

1. experience of qigong-related practice in the past 5 years;
2. reporting regular medication use that directly modulates immune system functioning (e.g., steroids, cytokine inhibitors, high levels of non-steroidal anti-inflammatory medication, chemotherapy, etc.) or sedates the nervous system (e.g., benzodiazepines, anti-epileptics, tranquilizers, etc.) or alters heart rate (e.g., beta blockers, calcium channel blocker, stimulants, etc.);
3. self-reported illicit drug use in the past 3 months or substance dependence over the past month (e.g., alcohol binge drinking 2+ days/week, using tobacco or nicotine products 5+ days/week, cannabis and related products 2+ days/week, etc.);
4. physical impairment that does not allow them to stand for 30 mins (e.g., severe obesity, need wheel-chair or equipment to assist with walking, recent injury that limits standing, etc.), and
5. severe mental health conditions that could prevent regular practice (e.g., hospitalized in the past 12 months for mental health condition).

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-08-29 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Increased heart rate variability | Day 1 in-person session, baseline T1 (before the intervention), the end of three-week intensive practice (T2), the end of the 3-month intervention (T3), the 6-month follow-up (T4), and the 12-month follow-up (T5).
  HRV will be collected using the H10 wear link and chest band (Polar Electro, Kempele, Finland) during several study activities, including 5 minutes of normal breathing at rest, a 5-minute paced-breathing task and during the 30-min intervention practice period. The normal and paced breathing assessments will occur at all data collection visits to estimate basal autonomic nervous system functioning.
Decreased inflammatory biomarker CRP | baseline T1 (before the intervention), the end of three-week intensive practice (T2), the end of the 3-month intervention (T3), the 6-month follow-up (T4), and the 12-month follow-up (T5).
  Saliva will be collected via approved methods (IBC BIO-23-0032). Salivary inflammatory biomarkers will be assessed in-house at the Biobehavioral Core Lab. Salivary C-reactive protein (sCRP) will be quantified using commercially available enzyme immunoassays according to manufacturer instructions. CRP is a protein produced by the liver in response to the cell mediated biomarker cytokines.
Decreased perceived stress | baseline T1 (before the intervention), the end of three-week intensive practice (T2), the end of the 3-month intervention (T3), the 6-month follow-up (T4), and the 12-month follow-up (T5).
  The 4-item Perceived Stress Scale measured on visual analogue ranging from 0 to 100, higher scores suggesting worse outcome.
Increased resilience | baseline T1 (before the intervention), the end of three-week intensive practice (T2), the end of the 3-month intervention (T3), the 6-month follow-up (T4), and the 12-month follow-up (T5).
  Brief Resilience Scale measured on visual analogue ranging from 0 to 100, higher scores suggesting better outcome.
Decreased fatigue | baseline T1 (before the intervention), the end of three-week intensive practice (T2), the end of the 3-month intervention (T3), the 6-month follow-up (T4), and the 12-month follow-up (T5).
  The 10-item Fatigue Assessment Scale measured on visual analogue ranging from 0 to 100, higher scores suggesting worse outcome.
Increased vitality | baseline T1 (before the intervention), the end of three-week intensive practice (T2), the end of the 3-month intervention (T3), the 6-month follow-up (T4), and the 12-month follow-up (T5).
  The 6-item Subjective Vitality Scale measured on visual analogue ranging from 0 to 100, higher scores suggesting better outcome.
Increased mystical experiences | baseline T1 (before the intervention), the end of three-week intensive practice (T2), the end of the 3-month intervention (T3), the 6-month follow-up (T4), and the 12-month follow-up (T5).
  The brief 8-item Mysticism Scale measured on visual analogue ranging from 0 to 100, higher scores suggesting better outcome.
Increased overall human flourishing | baseline T1 (before the intervention), the end of three-week intensive practice (T2), the end of the 3-month intervention (T3), the 6-month follow-up (T4), and the 12-month follow-up (T5).
  The 12-item Human Flourishing Measure measured on visual analogue ranging from 0 to 100, higher scores suggesting better outcome.

SECONDARY OUTCOMES:
Decreased inflammatory biomarker cytokine IL-1ß | baseline T1 (before the intervention), the end of three-week intensive practice (T2), the end of the 3-month intervention (T3), the 6-month follow-up (T4), and the 12-month follow-up (T5).
  Saliva will be collected via approved methods (IBC BIO-23-0032). Salivary inflammatory biomarkers will be assessed in-house at the Biobehavioral Core Lab. Plates will be read with a QuickPlex SQ 120 imager and data analyzed using the Discovery Workbench 4.0 for cytokines, including Interleukin (IL)-1ß.
Decreased inflammatory biomarker cytokine IL-6 | baseline T1 (before the intervention), the end of three-week intensive practice (T2), the end of the 3-month intervention (T3), the 6-month follow-up (T4), and the 12-month follow-up (T5).
  Saliva will be collected via approved methods (IBC BIO-23-0032). Salivary inflammatory biomarkers will be assessed in-house at the Biobehavioral Core Lab. Plates will be read with a QuickPlex SQ 120 imager and data analyzed using the Discovery Workbench 4.0 for cytokines, including Interleukin (IL)-6.
Decreased inflammatory biomarker cytokine TNF-a | baseline T1 (before the intervention), the end of three-week intensive practice (T2), the end of the 3-month intervention (T3), the 6-month follow-up (T4), and the 12-month follow-up (T5).
  Saliva will be collected via approved methods (IBC BIO-23-0032). Salivary inflammatory biomarkers will be assessed in-house at the Biobehavioral Core Lab. Plates will be read with a QuickPlex SQ 120 imager and data analyzed using the Discovery Workbench 4.0 for cytokines, including TNF-a.
Increased interoceptive awareness | baseline T1 (before the intervention), the end of three-week intensive practice (T2), the end of the 3-month intervention (T3), the 6-month follow-up (T4), and the 12-month follow-up (T5).
  The subscales Noticing, Attention Regulation, Emotional Awareness, Self-Regulation, and Body Listening of Multidimensional Assessment of Interoceptive Awareness - 2 measured on visual analogue ranging from 0 to 100, higher scores suggesting better outcome.
Reduced depression | baseline T1 (before the intervention), the end of three-week intensive practice (T2), the end of the 3-month intervention (T3), the 6-month follow-up (T4), and the 12-month follow-up (T5).
  Patient-Reported Outcomes Measurement Information System measured on visual analogue ranging from 0 to 100, higher scores suggesting worse outcome.
Reduced anxiety | baseline T1 (before the intervention), the end of three-week intensive practice (T2), the end of the 3-month intervention (T3), the 6-month follow-up (T4), and the 12-month follow-up (T5).
  Patient-Reported Outcomes Measurement Information System measured on visual analogue ranging from 0 to 100, higher scores suggesting worse outcome.

OTHER OUTCOMES:
Psychological Insight | baseline T1 (before the intervention), the end of three-week intensive practice (T2), the end of the 3-month intervention (T3), the 6-month follow-up (T4), and the 12-month follow-up (T5).
  The 14-item subscale Avoidance and Maladaptive Patterns Insights of the Psychological Insight measured on visual analogue ranging from 0 to 100, higher scores suggesting better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- University of North Carolina at Charlotte, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Funding Information — http://doi.org/10.54224/32539